CLINICAL TRIAL: NCT04508530
Title: A Superiority Phase III Study To Compare The Effect of Panzyga Versus Placebo in Patients With Pediatric Acute-onset Neuropsychiatric Syndrome (PANS/PANDAS)
Brief Title: Phase III Study To Compare The Effect of Panzyga Versus Placebo in Patients With Pediatric Acute-onset Neuropsychiatric Syndrome (PANS/PANDAS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NGAM-13
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Acute-Onset Neuropsychiatric Syndrome
MeSH Terms: conditions — Pediatric acute-onset neuropsychiatric syndrome | interventions — Panzyga

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Panzyga (Experimental): Panzyga 10% IVIG
  Interventions: Biological: Panzyga
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Panzyga — Panzyga 10% IVIG
  Arms: Panzyga
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A Superiority Study To Compare The Effect of Panzyga Versus Placebo in Patients with Pediatric Acute-onset Neuropsychiatric Syndrome

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥6 to ≤17 years of age.
2. Confirmed diagnosis of moderate to severe PANS with prominent and stable obsessive-compulsive disorder (OCD) symptoms (i.e. Clinical Global Impression (CGI)-Severity-OCD rating of ≥ 4 or higher on 2 ratings without a change of more than 1 unit between measurements) based on the following criteria:

   1. Abrupt dramatic onset of OCD meeting DSM-5 diagnostic criteria for OCD as confirmed by the MINI-KID-7
   2. Concurrent presence of additional neuropsychiatric symptoms, with similarly severe and acute onset, from at least two of the following seven categories, that are not better explained by a known neurologic or medical disorder, such as Sydenham chorea (SC), systemic lupus erythematosus, Tourette disorder, or other:

      * Anxiety (particularly, separation anxiety)
      * Emotional lability (extreme mood swings) and/or depression
      * Irritability, aggression and/or severely oppositional behaviors
      * Behavioral (developmental) regression (examples, talking baby talk,throwing temper tantrums, etc.)
      * Deterioration in school performance
      * Sensory or motor abnormalities
      * Somatic signs and symptoms, including sleep disturbances, bed wetting or urinary frequency
3. Signed informed consent of patient's legal representative(s)/guardians(s). If patients are old enough to understand the risks and benefits of the study (as determined by each institution), they should provide written assent/consent.
4. Legal representative(s)/guardians(s) must be capable of understanding and complying with the relevant aspects of the study protocol.

Patients who will additionally meet the following optional inclusion criteria will be identified as patients with Pediatric autoimmune neuropsychiatric disorders associated with streptococcal infection (PANDAS):

1. An episodic (relapsing-remitting) course of symptom severity
2. Temporal association between symptoms onset or exacerbation and infections with group A streptococcal infection (GAS, positive throat culture and/or anti-GAS antibody titers)

Exclusion Criteria

1. Onset of current PANS episode more than 12 months prior to first investigational medicinal product (IMP) treatment.
2. a. In patients with relapsing episodes: Onset of initial PANS episode more than 24 months prior to first IMP treatment.

   b. In patients with relapsing episodes: Absence of significant improvement and stabilization between the episodes according to investigator's judgment.
3. Contraindication to receiving intravenous immunoglobulin (IVIG), including:

   1. History of severe hypersensitivity, e.g. anaphylaxis or severe systemic response, to immunoglobulin, blood or plasma derived products, or any component of Panzyga.
   2. Immunoglobulin (Ig) A deficiency with antibodies to IgA (<7 mg/dL).
   3. Hyperviscosity syndromes or known or suspected hypercoagulable conditions as inferred from clinical history, which can increase risks of thrombosis associated with IVIG administration.
   4. History of arterial or venous thrombotic or thromboembolic events (TEEs) within the last year prior to Baseline. History of acquired or inherited thrombophilia any time prior to Baseline.
   5. Need for live virus vaccine within three months after receiving study drug.
   6. Renal dysfunction (creatinine >120 µmol/L or 1.36 mg/dL), history of renal dysfunction, or known risk factor for renal dysfunction (chronic renal insufficiency, diabetes mellitus, taking known nephrotoxic medication). For Italy, estimated glomerular filtration rate (eGFR) needs to be calculated with the 2009 Schwartz equation (eGFR = k * height/Serum creatinine (Scr), where k is 0.413) [2]. eGFR must not be below 30.
4. Severely restricted food intake likely to require parenteral nutrition, and <5th percentile BMI-for-age (BMI Percentile Calculator for Child and Teen based on Centers for Disease Control and Prevention growth charts for children and teens ages 2 through 19 years)
5. Body mass index ≥ 40 kg/m2
6. Presence of symptoms consistent with autism or schizophrenia, bipolar disorder, or other psychotic disorder (unless psychotic symptoms have onset coincident with PANS).
7. Presence of serious or unstable medical illness, psychiatric (e.g. high suicide risk) or behavioral symptoms that would make participation unsafe or study procedures too difficult to tolerate.
8. Treatment with systemic corticosteroids within eight weeks before randomization.
9. Treatment with NSAIDs within five days before randomization.
10. Treatment with melatonin within one week before randomization
11. History of rheumatic fever, including SC (neurological manifestation).
12. Past treatment of neuropsychiatric symptoms with immunomodulatory therapy (such as IVIG, rituximab or mycophenolate mofetil) or plasmapheresis.
13. Initiation of cognitive behavioral therapy (CBT) within eight weeks before randomization.
14. Start of treatment or change in dosing with selective serotonin reuptake inhibitors [SSRIs] within eight weeks before randomization.
15. Treatment with alpha-2 agonists or antipsychotics within eight weeks before randomization.
16. Start of treatment or change in dosing with stimulants (Methylphenidate, Amphetamine and similar products) for Attention-Deficit Hyperactivity Disorder (ADHD) within four weeks prior to randomization.
17. Active use of tetrahydrocannabinol (THC) containing agents within four weeks prior to enrollment or during the trial. Use of cannabidiol- (CBD) / cannabimovone- (CBM) containing agents without THC is allowed if started more than eight weeks before enrollment in a stable dose/frequency.
18. Use of antibiotics or antiviral drugs at therapeutic dose within one week before randomization. Use of antibiotics at a prophylactic dose is allowed if started at least four weeks before randomization (Section 4.2).
19. Severe liver disease (alanine aminotransferase [ALT] three times above normal value).
20. Known hepatitis B, hepatitis C or HIV infection as per patient medical history.
21. Cardiac insufficiency (New York Heart Association [NYHA] classification III-IV), cardiomyopathy, significant cardiac dysrhythmia requiring treatment.
22. Medical conditions with symptoms and effects that could alter protein catabolism and/or IgG utilization (e.g. protein-losing enteropathies, nephrotic syndrome).
23. Pregnant and/or lactating women.
24. Female patients of childbearing potential unwilling to use a protocol-required method of contraception (as per protocol Section 7.3.9 b) from Screening throughout the study treatment period and for four weeks following the last dose of study drug. A woman of childbearing potential is defined as a fertile woman or adolescent, from the beginning of menstruation, unless permanently sterile.
25. Participation in another interventional clinical trial that is either blinded or involves an investigational (not approved) product within three months before Baseline or during the course of the clinical study. Participation in observational clinical trials or open-label trials involving an approved product may be permitted after consultation with the medical monitor.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-10-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (7):
  - Octapharma Research Site, Tucson, Arizona
  - Octapharma Research Site, Little Rock, Arkansas
  - Octapharma Research Site, Los Angeles, California
  - Octapharma Research Site, Palo Alto, California
  - Octapharma Research Site, Centennial, Colorado
  - Octapharma Research Site, Boston, Massachusetts
  - Octapharma Research Site, Lebanon, New Hampshire
- Italy (2):
  - Octapharma Research Site, Genova
  - Octapharma Research Site, Roma
- Sweden (2):
  - Octapharma Research Site, Gothenburg
  - Octapharma Research Site, Stockholm

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo - Panzyga: Placebo until week 9 - Panzyga 10% (IVIG) until week 18
- Panzyga - Placebo: Panzyga 10% (IVIG) until week 9 - placebo until week 18
Period: First Intervention (Week 1-9)
Arm/Group | Placebo - Panzyga | Panzyga - Placebo
Started | 37 | 34
Completed | 36 | 28
Not Completed | 1 | 6
Period: Second Intervention (Week 10-18)
Arm/Group | Placebo - Panzyga | Panzyga - Placebo
Started | 36 | 28
Completed | 32 | 28
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo - Panzyga | Panzyga - Placebo | Total
Number analyzed (Participants) | 37 | 34 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 37 | 34 | 71
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.8 (2.95) | 9.3 (2.52) | 9.5 (2.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 11 | 30
  Male | 18 | 23 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 32 | 30 | 62
  Unknown or Not Reported | 0 | 1 | 1
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 18.99 (3.980) | 19.18 (4.755) | 19.08 (4.337)

OUTCOME MEASURES:

1. Secondary Outcome: Percentage Change in Total CY-BOCS Score From Week 9 to Week 18 Within the (Panzyga - Placebo) Treatment Sequence Group
Description: The CY-BOCS scores at the end of the follow up period were compared with the Week 9 scores to examine the durability of any clinical benefit following Panzyga treatment in the first 9-week treatment period and whether there was any worsening after crossing over to placebo treatment.
  The CY-BOCS scale score is a clinician-rated, semi-structured interview for rating the presence or absence, as well as the severity of obsessive-compulsive symptoms. The CY-BOCS yields a total obsession score, a total compulsion score and combined total score (minimum total CY-BOCS score=0, maximum total CY-BOCS score=40).
  The mean percentage change of the total CY-BOCS score at Week 18 to the Week 9 score was calculated within the (Panzyga - Placebo) treatment sequence group. A value of 0 means there was no change from Week 9 to Week 18. Negative values indicate a worse outcome. Positive values mean a better outcome.
Time Frame: 9 Weeks (Week 9 to Week 18)
Measure: Mean (Standard Deviation); unit: Percentage Change at Week 18 to Week 9
Groups:
- Panzyga - Placebo: Panzyga 10% (IVIG) Baseline to Week 9 - Placebo (0.9% w/v sodium chloride) Week 9 to Week 18
Arm/Group | Panzyga - Placebo
Number analyzed (Participants) | 25
Percentage Change at Week 18 to Week 9 | 29.4 (42.84)

2. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I) Score at Week 9
Description: The CGI-I rating scale was used to assess behavioral changes in PANS patients. The Clinical Global Impression - Improvement scale (CGI-I) is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention and is rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. The mean CGI-I scores at Week 9 were compared between Panzyga and placebo treatment.
Time Frame: 9 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo - Panzyga: Placebo (0.9% w/v sodium chloride) until week 9 - Panzyga 10% (IVIG) until week 18
- Panzyga - Placebo: Panzyga 10% (IVIG) until week 9 - placebo (0.9% w/v sodium chloride) until week 18
Arm/Group | Placebo - Panzyga | Panzyga - Placebo
Number analyzed (Participants) | 36 | 29
score on a scale | 3.3 (1.19) | 2.6 (1.32)
Statistical Analysis 1: Comparison: Placebo - Panzyga vs Panzyga - Placebo; Test type: Superiority; p = 0.00855, Mixed Models Analysis; Least Squares Mean Difference = 1.1, 5% CI 2-sided [0.2 to 2.0]

3. Primary Outcome: Percentage Change in CY-BOCS Score From Baseline to Week 9
Description: The primary endpoint of this study was the percentage change of neuropsychiatric symptomatology and behavior in PANS patients determined by clinician-rated Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) score.
  The CY-BOCS scale score is a clinician-rated, semi-structured interview for rating the presence or absence, as well as the severity of obsessive-compulsive symptoms. The CY-BOCS yields a total obsession score, a total compulsion score and combined total score (minimum total CY-BOCS score=0, maximum total CY-BOCS score=40).
  The mean percentage change in the total CY-BOCS score from Baseline to Week 9 was calculated and compared between Panzyga and Placebo treatment to demonstrate superiority. A value of 0 means there was no change from baseline to week 9. Negative values indicate a worse outcome. Positive values mean a better outcome.
Time Frame: 9 Weeks
Measure: Mean (Standard Deviation); unit: Percentage Change at Week 9 to Baseline
Arm/Group | Placebo - Panzyga | Panzyga - Placebo
Number analyzed (Participants) | 36 | 29
Percentage Change at Week 9 to Baseline | 12.1 (68.39) | 31.1 (40.68)
Statistical Analysis 1: Comparison: Placebo - Panzyga vs Panzyga - Placebo; Test type: Superiority; p = 0.0718, t-test, 1 sided; Mean Difference (Net) = -19.0, 2.5% CI 1-sided [upper limit 6.7]

4. Other Pre Specified Outcome: Patients With PANS Improvement From Baseline to Week 9
Description: The percentage of patients who showed PANS improvement was measured by Clinical Global Impression - Improvement (CGI-I) rating.
  "The Clinical Global Impression - Improvement is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a Baseline state at the beginning of the intervention and is rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse." PANS improvement was defined as a CGI-I rating of 1 (Very much Improved), 2 (Much improved), or 3 (Minimally Improved). The percentages of improved patients at Week 9 were compared to baseline between Panzyga and placebo treatment.
Time Frame: 9 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo - Panzyga | Panzyga - Placebo
Number analyzed (Participants) | 36 | 29
Participants
  PANS Improvement YES | 19 | 24
  PANS Improvement NO | 17 | 5
Statistical Analysis 1: Comparison: Placebo - Panzyga vs Panzyga - Placebo; Test type: Superiority; p = 0.0111, Chi-squared

ADVERSE EVENTS:
Time Frame: 18 weeks
Groups:
- Panzyga: Panzyga 10% (IVIG)
- Placebo: Placebo (0.9% w/v sodium chloride)
- Placebo After Panzyga: Placebo after Panzyga 10% (IVIG)
Arm/Group | Panzyga | Placebo | Placebo After Panzyga
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/37 | 0/27
Serious Adverse Events (participants affected / at risk) | 5/70 | 1/37 | 0/27
Other Adverse Events (participants affected / at risk) | 64/70 | 26/37 | 19/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panzyga (N=70) | Placebo (N=37) | Placebo After Panzyga (N=27)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Obsessive-compulsive Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panzyga (N=70) | Placebo (N=37) | Placebo After Panzyga (N=27)
Nausea (Gastrointestinal disorders) | 34 (54) | 8 (11) | 2 (2)
Vomiting (Gastrointestinal disorders) | 32 (52) | 2 (2) | 2 (3)
Upper Abdominal Pain (Gastrointestinal disorders) | 12 (17) | 3 (5) | 2 (2)
Headache (Nervous system disorders) | 57 (137) | 11 (18) | 3 (4)
Pyrexia (General disorders) | 30 (41) | 8 (9) | 3 (3)
Chills (General disorders) | 5 (6) | 3 (3) | 0 (0)
Fatigue (General disorders) | 8 (10) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (9) | 1 (1)
Coombs direct test positive (Investigations) | 7 (11) | 0 (0) | 1 (2)
Haemoglobin Decreased (Investigations) | 7 (8) | 1 (2) | 0 (0)
Behaviorous Disorders (Psychiatric disorders) | 1 (1) | 1 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 2 (2) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 4 (5) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 5 (6) | 2 (3) | 0 (0)
Pain (General disorders) | 4 (4) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (4) | 3 (3) | 2 (3)
COVID-19 (Infections and infestations) | 4 (4) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 1 (1)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Peripheral Swelling (General disorders) | 0 (0) | 2 (2) | 1 (1)
Free haemoglobin present (Investigations) | 0 (0) | 2 (2) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT04508530/Prot_002.pdf
  • Statistical Analysis Plan (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT04508530/SAP_003.pdf